CLINICAL TRIAL: NCT07026305
Title: Non-inferiority of Osseous Decompression of the Lumbar Canal Until Normalization of Epidural Pressure Compared to Conventional Open Laminectomy in Patients With Symptomatic Lumbar Spinal Stenosis.
Brief Title: Is it Really Necessary Going All Over the Top in Patients With Symptomatic Lumbar Spinal Stenosis?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Hospital San Carlos, Madrid (Other); FUNDACION PARA LA INVESTIGACION HOSPITAL CLINICO SAN CARLOS (Other)
Responsible Party: Principal Investigator, Juan Pablo Castaño Montoya, M.D., M.Sc., Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24/605-EC-X_Tesis
Record Dates: First submitted 2025-06-05; First posted 2025-06-18 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Lumbar Canal Stenosis; Lumbar Spinal Stenosis; Lumbar Spinal Stenosis (LSS)
Keywords: lumbar canal stenosis; spinal epidural pressure; lumbar spinal stenosis; LSS
MeSH Terms: conditions — Spinal Stenosis | interventions — Laminectomy

STUDY DESIGN:
Intervention Model Description: This is a non-inferiority, controlled, randomized, single-blind clinical trial comparing the effectiveness of full lumbar canal bony decompression up to normalization of epidural pressure versus open laminectomy in patients with symptomatic lumbar canal stenosis.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pressure-guided laminectomy (PGL) (Experimental): Osseous resection of the lamina and ligamentum flavum until the epidural pressure reaches a normal value at the stenotic segment.
  Interventions: Procedure: Pressure-guided laminectomy (PGL)
- Non-pressure-guided laminectomy (NPGL) (Active Comparator): Complete resection of both the lamina and the ligamentum flavum at the stenotic segment.
  Interventions: Procedure: Laminectomy without pressure guidance (LWPG)

INTERVENTIONS:
Procedure: Pressure-guided laminectomy (PGL) — Osseous resection of the lamina and ligamentum flavum until the epidural pressure reaches a normal value at the stenotic segment.
  Arms: Pressure-guided laminectomy (PGL)
Procedure: Laminectomy without pressure guidance (LWPG) — Complete resection of both the lamina and the ligamentum flavum at the stenotic segment.
  Arms: Non-pressure-guided laminectomy (NPGL)

SUMMARY:
The goal of this clinical trial is to evaluate the theory of epidural pressure by comparing a surgical procedure that aims to perform less bone resection compared to conventional surgery in patients with lumbar spinal stenosis.

The main questions it aims to answer is:

Is bony decompression of the lumbar canal performed until normalization of epidural pressure not inferior to conventional surgery in achieving clinical improvement in patients with symptomatic lumbar canal stenosis?

Researchers will:

Compare conventional open laminectomy to bony decompression of the lumbar canal until normalization of epidural pressure is achieved.

Participants will:

* Be randomized to one of the two surgical interventions: laminectomy guided by epidural pressure measure or conventional laminectomy.
* Visit the clinic for checkups and tests until 1 year of follow-up.

DETAILED DESCRIPTION:
This is a non-inferiority, controlled, randomized, single-blind clinical trial comparing the effectiveness of full lumbar canal bony decompression up to normalization of epidural pressure versus open laminectomy in patients with symptomatic lumbar canal stenosis. The study will not involve any medical industry sponsorship.

Surgical intervention decisions will be made by a single neurosurgeon at Hospital Clínico San Carlos, based on clinical scales and imaging as specified in the inclusion criteria. After the patient signs the informed consent form and is placed on the surgical waiting list, they will be randomized in a 1:1 ratio (simple randomization implemented via SPSS software). Baseline clinical scales will be administered (Zurich Claudication Questionnaire, ZCQ; Numeric Pain Rating Scale, NPRS; Oswestry Disability Index, ODI; Japanese Orthopaedic Association Back Pain Evaluation Questionnaire, JOABPEQ) to establish the patient's baseline status. The patient will remain blinded to the assigned intervention group.

Study Interventions:

* Pressure-guided laminectomy (PGL): An open laminectomy with complete decompression of the posterior elements. This is defined as the classic technique. After muscle dissection, a Codman microsensor (Integra LifeSciences) is inserted into the epidural space under direct visualization, performing careful dissection of the inferior aspect of the ligamentum flavum on the right hemilamina to obtain the patient's baseline epidural pressure. The sensor is then removed, and resection of the spinous process, supraspinous and interspinous ligaments, bilateral hemilaminae, and ligamentum flavum is performed until an adequate decompression of the thecal sac is achieved.
* Non-pressure-guided laminectomy (NPGL): After muscle dissection, the Codman microsensor is inserted into the epidural space as described above. The patient's baseline epidural pressure is recorded, and then bony decompression is initiated using the "unilateral laminotomy for bilateral decompression" technique from the left side, continuing until the epidural pressure decreases to 10 mmHg, a value established as the median within normal range.

The CODMAN Microsensor pressure catheter (Integra LifeSciences) is a transducer with a distal strain gauge that records pressure changes in a given medium. Its proximal end has an electrical connector that must be attached to the ICP Express monitor. This particular microsensor model was chosen due to its availability in the operating room inventory and because it has been used in previous studies published in the scientific literature.

All surgeries will be performed by a single neurosurgeon at Hospital Clínico San Carlos. Patients will be evaluated two weeks after surgery, at which time clinical scales will be applied and the surgical wound will be checked. Subsequently, patients will be evaluated at 3 and 6 months postoperatively via telephone follow-up, and at 12 months with an in-person visit, during which clinical outcome scales will be administered.

Additionally, a lumbosacral MRI will be obtained 3 months after surgery to qualitatively assess the degree of decompression achieved in each patient.

Sociodemographic data and clinical outcome variables will be collected during the preoperative consultation and at the follow-up visits at 1, 3, 6, and 12 months post-surgery. Imaging data will be collected from the patient's preoperative lumbar spine MRI (baseline) and from the lumbar MRI obtained 3 months postoperatively. T2-weighted axial sequences will be used to qualitatively assess the extent of bony decompression.

The database generated for the study will not contain any patient identifiers, thus maintaining confidentiality of patient identity. Study data will be recorded in a de-identified manner linked to a unique code per patient, such that only the researcher can associate these data with an individual medical record. Access to participants' clinical documentation will be limited to the investigators and personnel responsible for data quality assurance and analysis.

All procedures will adhere to Regulation (EU) 2016/679 of the European Parliament and of the Council of 27 April 2016 (General Data Protection Regulation), and to Spanish Organic Law 3/2018 of December 5 on Personal Data Protection and Guarantee of Digital Rights (LOPDGDD). The entity responsible for data processing is Hospital Clínico San Carlos, whose Data Protection Officer is the DPO Committee of the Regional Health Authority of the Community of Madrid. This entity will handle data for the purposes outlined in this document.

Personal data, including health data, will be retained for the duration of the project and up to three years after its conclusion. Patients may exercise their rights of access and rectification of data, as well as the right to restrict data processing and to request a copy of their data or transfer of their data to a third party.

Descriptive statistics will be used to summarize the demographic and clinical data. Quantitative variables will be summarized by their mean and standard deviation (SD) if normally distributed. Quantitative variables with a skewed distribution will be summarized by median and interquartile range (IQR). Qualitative variables will be presented as frequency distributions.

No interim efficacy analysis will be performed.

Efficacy analysis will be conducted on both the Per-Protocol (PP) and Intention-to-Treat (ITT) populations. Safety analysis will be performed only on the ITT population. Data will be examined longitudinally, and the primary analysis will focus on differences in effectiveness between the two intervention modalities as measured by the ZCQ and the other clinical scales over time. Interaction terms between treatment group and time will also be included to explore whether effects differ across follow-up time points.

Non-inferiority efficacy analysis will be carried out using linear regression models with a one-sided α of 0.05 and using the non-inferiority margins. Multiple non-inferiority hypotheses will be tested (one for each clinical scale); adjustments for multiple comparisons will be applied to control the overall Type I error rate, progressively tightening the alpha for each additional hypothesis so that the study maintains the required overall error threshold.

In addition to unadjusted analyses, all analyses will be adjusted for potential confounding factors such as age, sex, and comorbidities using multiple linear regression.

For the safety analysis, any complications occurring during the study period will be analyzed. Their association with the type of intervention will be evaluated using logistic regression models. In this case, a two-sided α level of 0.05 will be considered.

All results from the analyses will be expressed as estimated mean effects with 95% confidence intervals, and these estimates will be compared against the non-inferiority margin to infer non-inferiority of the intervention. The analyses described above will be conducted using IBM SPSS Statistics v26 and R v4.4.1.

Resources for the Study

* Human resources: Neurosurgeon; Neurosurgery resident; Methodological research support unit (UAMI).
* Physical resources: Scheduled surgery operating room; Outpatient clinic office (with chair, desk, computer, and examination table); Data analysis room with computer.
* Specific materials: Intracranial pressure monitoring catheter (Codman); Intracranial pressure monitor.

Timeline The expected duration of the trial is 2 years, subdivided into a 12-month patient recruitment period and 1 year of follow-up.

Adverse Events It is the investigator's responsibility to detect and document any occurrence meeting the criteria and definition of an adverse event (AE). Adverse events will be reported as per the guidelines established by the CONSORT Statement for Randomized Trials of Nonpharmacologic Treatments: 2017 Update and Extension for Nonpharmacologic Trial Abstracts.

Ethical Considerations The trial will be conducted in accordance with the principles of the Declaration of Helsinki and the current legal regulations in Spain. It will commence only after obtaining approval from the relevant Research Ethics Committee (Comité Ético de Investigación Clínica, CEIC).

Plan for Dissemination of Results Upon completion of the study, publications will be prepared to disseminate the findings in national or international journals, and the results will also be presented at conferences. The principal investigator commits to complying with current Spanish legislation, which mandates the publication of all results (positive or negative) in scientific journals, including reference to the approving CEIC and the study's funding source.

ELIGIBILITY:
Inclusion Criteria:

* Surgical indication determined by:

  * Lower back pain and/or lower extremity pain for more than 3 months.
  * Pain refractory to conservative medical management (analgesics, physical therapy, epidural block).
  * Clinical criterion of neurogenic claudication defined as a score ≥11 on the N-CLASS scale.
  * Preoperative magnetic resonance imaging (MRI) showing lumbar canal stenosis.
* Patient consents to the proposed surgical intervention.
* Patient agrees to participate in the study by signing the informed consent form.

Exclusion Criteria:

* Foraminal or lateral recess stenosis.
* Symptomatic disc herniation at the segment to be treated.
* Spondylolisthesis > Grade I (Meyerding) (translation >25% of the vertebra) or spondylolysis.
* Radiological instability defined as >5 mm of anteroposterior translation on dynamic flexion-extension spine X-rays.
* Scoliosis with Cobb angle >30°.
* Compression fracture at the level to be treated.
* Prior surgery at the same segment to be treated.
* Prior infection at the segment to be treated.
* Contraindication for MRI.
* Diagnosis of major depressive disorder or dysthymia according to DSM-V criteria.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Zurich Claudication Questionnaire (ZCQ) - Symptom Severity subcategory. | At enrollment and at the follow-up visits at 1, 3, 6, and 12 months post-surgery.
  This scale consists of 7 items that evaluate the severity of symptoms over the last month on a numeric scale from 1 to 5, where 5 represents greater severity. A mean score of the items is calculated.

SECONDARY OUTCOMES:
Zurich Claudication Questionnaire (ZCQ) - Physical Function subcategory. | At enrollment and at the follow-up visits at 1, 3, 6, and 12 months post-surgery.
  Consists of 5 items evaluating functional impairment over the last month on a numeric scale from 1 to 4, where 4 represents greater disability. A mean score of the items is calculated.
Zurich Claudication Questionnaire (ZCQ) - Patient Satisfaction subcategory. | At enrollment and at the follow-up visits at 6 and 12 months post-surgery.
  Consists of 5 items, classified into 4 categories (from very satisfied to very dissatisfied), assessing overall outcome, pain relief, walking ability, ability to work or do house/garden chores, and strength and balance. This subcategory is assessed at 6 months and 1 year post-surgery.
Numeric Pain Rating Scale (NPRS). | At enrollment and at the follow-up visits at 1, 3, 6, and 12 months post-surgery.
  A pain measurement scale where patients rate their pain on an 11-point scale from 0 to 10, with 0 (far left) representing "no pain" and 10 (far right) representing "worst imaginable pain." This will be evaluated for both lower extremity symptoms (NPRS for legs) and for lower back/gluteal pain (NPRS for back or buttock).
Oswestry Disability Index (ODI). | At enrollment and at the follow-up visits at 1, 3, 6, and 12 months post-surgery.
  Assesses disability associated with pain across 10 items, each scored from 0 (no disability) to 5 (severely affected). The result is a percentage score calculated as the sum of item scores divided by the total possible points, multiplied by 100. Disability is classified as minimal (0-20%), moderate (21-40%), severe (41-60%), crippled (61-80%), or bed-bound/exaggeration (>80%).
Japanese Orthopaedic Association Back Pain Evaluation Questionnaire (JOABPEQ). | At enrollment and at the follow-up visits at 1, 3, 6, and 12 months post-surgery.
  Covers five domains-pain-related disorders, lumbar spine dysfunction, gait disturbance, social life dysfunction, and psychological disorders. JOABPEQ scores range from 0 to 100, with higher scores indicating better health status.
Surgical complications. | From enrollment to the end of the follow-up at 1 year.
  Any perioperative or postoperative complication related to the surgery.
Surgical re-intervention. | From enrollment to the end of the follow-up at 1 year.
  Any subsequent surgical procedure required on the same spinal level during the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Juan P Castaño-Montoya, M.D.,M.Sc., Principal Investigator — Universidad Complutense de Madrid; Angela M Carrascosa-Granada, M.D.,M.Sc.,Ph.D., Study Director — Universidad Complutense de Madrid
Locations (1):
- Hospital Clínico San Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
At this time, a decision has not yet been made regarding the sharing of individual participant data (IPD). The research team is currently evaluating the ethical, legal, and logistical considerations involved, including participant privacy concerns and data governance policies. A final decision will be made upon completion of the study and in accordance with institutional guidelines and applicable regulations.

REFERENCES:
- [Background] Zhang C, Chen L, Li J, Huang D, Zhang W, Lin J. Should Posterior Midline Structures Be Preserved in Decompression Surgery for Lumbar Spinal Stenosis?: A Systematic Review and Meta-analysis. Clin Spine Surg. 2022 Oct 1;35(8):341-349. doi: 10.1097/BSD.0000000000001268. Epub 2021 Oct 28. PMID 34711752
- [Background] Soliman MAR, Ali A. Decompression of lumbar canal stenosis with a bilateral interlaminar versus classic laminectomy technique: a prospective randomized study. Neurosurg Focus. 2019 May 1;46(5):E3. doi: 10.3171/2019.2.FOCUS18725. PMID 31042649
- [Background] Boukebir MA, Berlin CD, Navarro-Ramirez R, Heiland T, Scholler K, Rawanduzy C, Kirnaz S, Jada A, Hartl R. Ten-Step Minimally Invasive Spine Lumbar Decompression and Dural Repair Through Tubular Retractors. Oper Neurosurg. 2017 Apr 1;13(2):232-245. doi: 10.1227/NEU.0000000000001407. PMID 28927213
- [Background] Takahashi K, Miyazaki T, Takino T, Matsui T, Tomita K. Epidural pressure measurements. Relationship between epidural pressure and posture in patients with lumbar spinal stenosis. Spine (Phila Pa 1976). 1995 Mar 15;20(6):650-3. PMID 7604339
- [Background] Barz T, Melloh M, Staub LP, Lord SJ, Lange J, Merk HR. Increased intraoperative epidural pressure in lumbar spinal stenosis patients with a positive nerve root sedimentation sign. Eur Spine J. 2014 May;23(5):985-90. doi: 10.1007/s00586-013-3071-3. Epub 2013 Oct 29. PMID 24166020
- [Background] Takahashi K, Kagechika K, Takino T, Matsui T, Miyazaki T, Shima I. Changes in epidural pressure during walking in patients with lumbar spinal stenosis. Spine (Phila Pa 1976). 1995 Dec 15;20(24):2746-9. doi: 10.1097/00007632-199512150-00017. PMID 8747254
- [Background] Hermansen E, Myklebust TA, Weber C, Brisby H, Austevoll IM, Hellum C, Storheim K, Aaen J, Banitalebi H, Brox JI, Grundnes O, Rekeland F, Solberg T, Franssen E, Indrekvam K. Postoperative Dural Sac Cross-Sectional Area as an Association for Outcome After Surgery for Lumbar Spinal Stenosis: Clinical and Radiological Results From the NORDSTEN-Spinal Stenosis Trial. Spine (Phila Pa 1976). 2023 May 15;48(10):688-694. doi: 10.1097/BRS.0000000000004565. Epub 2023 Feb 20. PMID 36809364
- [Background] Gupta S, Bansal T, Kashyap A, Sural S. Correlation between clinical scoring systems and quantitative MRI parameters in degenerative lumbar spinal stenosis. J Clin Orthop Trauma. 2022 Oct 20;35:102050. doi: 10.1016/j.jcot.2022.102050. eCollection 2022 Dec. PMID 36317084
- [Background] Boden SD, Davis DO, Dina TS, Patronas NJ, Wiesel SW. Abnormal magnetic-resonance scans of the lumbar spine in asymptomatic subjects. A prospective investigation. J Bone Joint Surg Am. 1990 Mar;72(3):403-8. PMID 2312537
- [Background] Suner HI, Castano JP, Vargas-Jimenez A, Wagner R, Mazzei AS, Velazquez W, Jorquera M, Sallabanda K, Barcia Albacar JA, Carrascosa-Granada A. Comparison of the Tubular Approach and Uniportal Interlaminar Full-Endoscopic Approach in the Treatment of Lumbar Spinal Stenosis: Our 3-Year Results. World Neurosurg. 2023 May;173:e148-e155. doi: 10.1016/j.wneu.2023.02.022. Epub 2023 Feb 10. PMID 36775236
- [Background] Carrascosa-Granada A, Velazquez W, Wagner R, Saab Mazzei A, Vargas-Jimenez A, Jorquera M, Albacar JAB, Sallabanda K. Comparative Study Between Uniportal Full-Endoscopic Interlaminar and Tubular Approach in the Treatment of Lumbar Spinal Stenosis: A Pilot Study. Global Spine J. 2020 Apr;10(2 Suppl):70S-78S. doi: 10.1177/2192568219878419. Epub 2020 May 28. PMID 32528810
- [Background] Chen X, Zheng Z, Lin J. Clinical Effectiveness of Conservative Treatments on Lumbar Spinal Stenosis: A Network Meta-Analysis. Front Pharmacol. 2022 Jun 6;13:859296. doi: 10.3389/fphar.2022.859296. eCollection 2022. PMID 35734403
- [Background] Chad DA. Lumbar spinal stenosis. Neurol Clin. 2007 May;25(2):407-18. doi: 10.1016/j.ncl.2007.01.003. PMID 17445736
- [Background] Kobayashi H, Sekiguchi M, Yonemoto K, Kakuma T, Tominaga R, Kato K, Watanabe K, Nikaido T, Otani K, Yabuki S, Kikuchi SI, Konno SI; DISTO project working group. Reference values of the Japanese Orthopaedic Association Back Pain Evaluation Questionnaire in patients with lumbar spinal stenosis and characteristics of deterioration of QOL: Lumbar Spinal Stenosis Diagnosis Support Tool: DISTO project. J Orthop Sci. 2019 Jul;24(4):584-589. doi: 10.1016/j.jos.2018.11.022. Epub 2019 Jan 5. PMID 30616940
- [Background] Katz JN, Zimmerman ZE, Mass H, Makhni MC. Diagnosis and Management of Lumbar Spinal Stenosis: A Review. JAMA. 2022 May 3;327(17):1688-1699. doi: 10.1001/jama.2022.5921. PMID 35503342

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-06-02): https://cdn.clinicaltrials.gov/large-docs/05/NCT07026305/Prot_SAP_ICF_000.pdf